CLINICAL TRIAL: NCT00065689
Title: High Intensity Light Therapy in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT000212-01A1 (NIH); SloaneP
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; light therapy; long-term care; depression; sleep; agitation
MeSH Terms: conditions — Alzheimer Disease; Dementia; Depression; Psychomotor Agitation

INTERVENTIONS:
Device: high-intensity light therapy

SUMMARY:
The purpose of this study is to determine whether bright light improves the sleep, mood, and behavior of persons with Alzheimer's disease and related dementias (AD) who live in long-term care settings and, if so, to determine the best timing for the light therapy. The light levels being used in the study have been shown to improve depression in persons with seasonal affective disorder (SAD) and to relieve sleep problems in persons with jet lag and other body rhythm disturbances. Because persons with AD often will not remain still in front of a fluorescent panel, this project has involved renovations in the study units that provide for even, regulated, high-intensity light in all public areas of the study settings.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of dementia
* Residence on study units

Exclusion criteria:

* Bipolar disorder
* Severe retinal (eye) disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107
Dates: Start 2003-03; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Philip D. Sloane, MD, MPH, Principal Investigator
Locations (1):
- John Umstead Hospital, Butner, North Carolina, United States